CLINICAL TRIAL: NCT03357224
Title: Phase II Trial of Atezolizumab (Anti-PD-L1) in the Treatment of Stage IIb-IV Mycosis Fungoides/Sezary Syndrome Patients Relapsed/Refractory After a Previous Systemic Treatment
Brief Title: PARCT: Trial of Atezolizumab in Relapsed/Refractory Cutaneous T Cell Lymphoma (CTCL)
Acronym: PARCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following an urgent safety measure due to toxicity recruitment has been closed prematurely.
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC 1652-CLTF
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides/Sezary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Atezolizumab (Experimental): The treatment will be given for a maximum of 1-year unless confirmed disease progression or unless other criteria for treatment discontinuation are met as specified in the protocol.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Patients will receive atezolizumab 1200 mg IV Q3w for 1 year.
  Other Names: Tecentriq

SUMMARY:
Trial assessing atezolizumab (anti-PD-L1) as treatment option for patients with mycosis fungoides/sezary syndrome having progressed under or after previous therapy

For this study, we invite patients suffering from mycosis fungoides and Sézary syndrome who have progressed after initial therapy or have failed to respond to previous therapy.

Mycosis fungoides and Sézary syndrome are cancers in which lymphocytes* become malignant (cancerous) and affect the skin. In mycosis fungoides, the disease is generally limited to the skin, and people develop flat or raised areas on their skin where the lymphocytes have accumulated. Sometimes even larger aggregations of lymphocytes occur in the skin or lymph nodes, resulting in tumors. In Sézary syndrome, the skin is often reddened or itchy, and some abnormal lymphocytes circulate in the blood.

* Lymphocytes are a type of immune cells that is made in the bone marrow and is found in the blood. Lymphocytes have a number of roles in the immune system, including the production of antibodies and other substances that fight infections and other diseases.

In standard practice, the disease will be treated with conventional chemotherapy that unfortunately has a limited lasting benefit. In this study, we want to see if a new treatment option can optimize and improve response and make benefit last as long as possible. This new treatment option is immunotherapy, using atezolizumab (Tecentriq).

Immunotherapy is a cancer treatment that uses antibodies made in the laboratory from a single type of immune system cell. These antibodies can identify substances on cancer cells or normal cells that may help cancer cell grow. The antibodies attach to the substances and kill the cancer cells, block their growth, or keep them from spreading. Atezolizumab blocks a protein called PD-L1 (programmed death-ligand 1) from binding to its receptor found on the surface of lymphocytes. It helps to restore the immune activity of the body against the cancer.

Atezolizumab is already used to treat adults with a cancer that affects the bladder and the urinary system, called urothelial carcinoma, and a cancer that affects the lungs, called non-small cell lung cancer.

In this trial, patients will receive atezolizumab for one year unless the tumor starts growing again or this is not considered suitable for them anymore or they wish to stop the treatment.

ELIGIBILITY:
Inclusion criteria

* Male or female patients with diagnosis of CTCL (mycosis fungoides or Sézary-Syndrome) tumor stage IIB to IVB
* Mandatory to ship tumor sample for evaluation of PD-L1 expression. A 4 mm formalin-fixed punch biopsy is recommended.
* Inadequate response or secondary treatment failure to at least 1 prior systemic therapy for CTCL according to treatment guidelines (e.g. INF-2α or bexarotene).
* Age ≥ 18 years old
* WHO performance status 0-1
* Adequate bone marrow and organ function prior to receiving the first dose of study treatment:
* Hemoglobin >10.0 g/dL (>100 g/L) or hematocrit >30% (>0.30 v/v);
* White blood cell count >3.0 x 109/L (>3000/mm3);
* Absolute neutrophil count of >1.5 x 109/L (>1500/mm3);
* Platelet count >100 x 109/L (>100,000/mm3);
* Estimated creatinine clearance >40 mL/min based on the Cockcroft Gault calculation or serum creatinine less than 1.5 times the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) values less than 2 times the upper limit of normal (ULN)
* Serum total bilirubin 1.5 ULN
* Patients with suspicion of Gilbert disease who have serum bilirubin level 3 x ULN may be enrolled.
* Clinically normal cardiac function based on 12 lead ECG without clinically relevant abnormalities and the institutional lower limit of normal for left ventricular ejection fraction as assessed either by multi-gated acquisition scan or cardiac ultrasound.
* Women of child bearing potential (WOCBP) must have a negative serum pregnancy test within 72 hours prior to the first dose of study treatment.

Note: women of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e. females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons.

* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 5 months after the last dose of treatment. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Such methods include:
* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
* Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
* Intrauterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomized partner
* Sexual abstinence (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient)
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment.
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion criteria

* Patients for whom only local therapy is indicated.
* Received chemotherapy or targeted small molecule therapy within 4 weeks prior to registration.
* Persistence of clinically relevant therapy-related toxicity from previous systemic treatment. Grade 1 or 2 adverse events (AEs) are acceptable.
* Received a T cell depleting antibody (e.g. Campath) within 3 months prior to the first dose of atezolizumab.
* Prior therapy with anti-PD1, anti-PD-L1, anti-PD-L2.
* History of other malignancy in the past 5 years with the exception of treated carcinoma in situ of the cervix and non-metastatic, non-melanoma skin cancer.
* Patients with known central nervous system (CNS) involvement with lymphoma.
* History of severe allergic anaphylactic reactions to chimeric, human or humanized antibodies, or fusion proteins.
* Known hypersensitivity to CHO cell products or any component of the atezolizumab formulation.
* History of any of the following cardiovascular conditions within 6 months prior to the first dose of study treatment:
* Unstable angina.
* Clinically significant cardiac arrhythmias.
* Myocardial infarction.
* Have current or recent (past 6 months) history of severe, progressive, or uncontrolled renal, hepatic, gastrointestinal, metabolic, endocrine, pulmonary, cardiovascular, or neurological disease.
* Severe infection within 4 weeks prior to registration, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Have active signs of disseminated herpes zoster or disseminated herpes simplex, or a recurrent (more than one episode of) localized, dermatomal herpes zoster.
* Administration of a live, attenuated vaccine within 4 weeks prior to Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study. Any live, attenuated vaccine (e.g. FluMist®) is prohibited while the patient is receiving atezolizumab and for a period of 5 months after discontinuation of atezolizumab. Inactivated influenza vaccines are allowed only during flu season.
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:
* Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
* Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
* Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
* Rash must cover 10% of body surface area
* Disease is well controlled at baseline and requires only low-potency topical corticosteroids
* No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12months
* Has a known history of HIV (test to be performed within 21 days of registration)
* Has known active Hepatitis B or Hepatitis C. Note: patient will be eligible if
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening . The HBV DNA test will be performed only for patients who have a positive total HBcAb test.
* Has immunodeficiency or on systemic steroid / immunosuppressive therapy within 7 days prior to the first dose of atezolizumab.

Note: systemic corticosteroids at doses ≤ 10 mg/day of prednisone or its equivalent is permitted

* Current or previous history of non-infectious pneumonitis requiring steroids, or pulmonary fibrosis.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation.
* Evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB).
* Regarding hematopoietic stem cell transplantation:
* Patients who had previously stem cell transplantation
* Patients that are waiting for stem cell transplantation
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

All eligibility criteria must be adhered to, in case of deviation discussion with Headquarters and study coordinator is mandatory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Best overall response (CR+PR) rate (EORTC-ISCL-USCLC criteria) | Up to maximum 1 year starting from patient registration
  Overall response rate is defined as the proportion of patients with global response score equal to CR or PR

SECONDARY OUTCOMES:
Progression free survival (EORTC-International Society of Cutaneous Lymphoma (ISCL)-United States Cutaneous Lymphoma Consortium (USCLC) criteria) | 6 months as of Last Patient In (LPI)
  From registration to progression
Overall survival (OS) | 5 years as of LPI based on the median overall survival
  Registration till the date of death from any cause
Duration of response | 6 months as of LPI
  From registration to progression
Time to response (CR/PR) | 6 months as of LPI
  From registration to progression
Time to next systemic treatment | 8 months as of LPI
  Time from the end of the current atezolizumab treatment until the time the next systemic treatment is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Stadler, Study Chair — Johannes Wesling Klinikum Minden - Minden, Germany; Robert Knobler, Study Chair — Medical University Vienna, General Hospital AKH - Vienna, Austria
Locations (2):
- Hospital Universitario 12 De Octubre, Madrid, Spain
- UniversitaetsSpital Zurich - Division of Dermatology, Zurich, Switzerland